CLINICAL TRIAL: NCT06112938
Title: Alternative Treatment Strategies for Stenotrophomonas Maltophilia Pneumonia
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 034.PHA.2022.A
Record Dates: First submitted 2022-10-21; First posted 2023-11-02 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Stenotrophomonas Maltophilia Infection
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Antibiotic — We aim to examine differences in clinical outcomes and failure rates between standard and alternative treatment strategies such as minocycline (or moxifloxacin, ciprofloxacin, ceftazidime) alone or in combination with TMP-SMX, alternative TMP-SMX dosing regimens, or variations in durations of therapy for the treatment of S. maltophilia infections within Methodist Health System (MHS).

SUMMARY:
Multi center, retrospective chart review of patients admitted to MHS hospitals from April 1, 2017 to March 31, 2022. Patients will be identified through the electronic medical record, and data from those that meet the study inclusion and exclusion criteria will be analyzed. Minimum inhibitory concentration (MIC) data will be interpreted per Clinical & Laboratory Standards Institute (CLSI) standards to determine local patterns of resistance. Multivariable logistic regression will be performed to determine predictors of mortality for S. maltophilia isolates.

DETAILED DESCRIPTION:
Stenotrophomonas maltophilia is an aerobic, non-fermenting, Gram-negative bacillus recognized by the World Health Organization as one of the leading multi-drug resistant nosocomial pathogens worldwide. The Investigators aim to examine differences in clinical outcomes and failure rates between standard and alternative treatment strategies such as minocycline (or moxifloxacin, ciprofloxacin, ceftazidime) alone or in combination with TMP-SMX, alternative TMP-SMX dosing regimens, or variations in durations of therapy for the treatment of S. maltophilia infections within Methodist Health System (MHS).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* S. maltophilia isolated on respiratory or blood culture

Exclusion Criteria:

* Those that do not meet the inclusion criteria outlined in Section 4.1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective chart review study limited to only patients meeting inclusion and exclusion criteria. We plan to conduct the retrospective chart review of all patients identified during the study period that meet the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
the difference in clinical failure rates between standard and alternative therapy | 30 days
  defined as meeting any of the following criteria: 1) isolation of S. maltophilia from a subsequently collected culture from the same site of index culture after at least 48 hours of therapy; 2) alteration of monotherapy after at least 48 hours of treatment for either an adverse event or concern for clinical failure; or 3) 30-day in-hospital all-cause mortality.

SECONDARY OUTCOMES:
Clinical outcomes such as ICU LOS | 30 days
  related/attributable mortality, and rates of serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Crotty, PharmD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No